CLINICAL TRIAL: NCT00965042
Title: Effect of Ceftobiprole on the Intestinal Human Microflora Following Multiple-dose Administration in Healthy Female and Male Subjects
Brief Title: Effect of Ceftobiprole on Human Intestinal Microflora
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR016306; BAC-1002 (Other: Basilea Internal Reference)
Record Dates: First submitted 2009-08-21; First posted 2009-08-25 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Antimicrobial Agent; Cephalosporins; Drug Resistance
Keywords: Ceftobiprole; ZEVTERA; ZEFTERA; Intestinal Microflora
MeSH Terms: interventions — ceftobiprole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceftobiprole (Experimental): Ceftobiprole 500 mg by 2 hour intravenous infusion every 8 hours for 7 days
  Interventions: Drug: Ceftobiprole

INTERVENTIONS:
Drug: Ceftobiprole — ceftobiprole 500 mg by intravenous infusion every 8 hours for 7 days

SUMMARY:
The purpose of the study is to investigate the effect of ceftobiprole treatment on intestinal microflora in healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label, single center study to investigate the effect on human intestinal microflora of multiple doses of ceftobiprole treatment administered at 8 hours intervals for 7 consecutive days. Careful investigation of the effect of Ceftobiprole treatment on the intestinal microflora is of importance since alteration of the intestinal microflora balance may facilitate colonization by pathogenic bacteria strains or enable microorganisms already present in the normal microflora to develop resistance. A total of 7 fecal samples will be collected on day 2, 4, 7, 10, 14 and 21 for determination of ceftobiprole concentration in fecal, intestinal microflora pattern and measuring the susceptibility for Ceftobiprole of isolated bacterial strains. A total of 13 plasma samples will be collected on day 1, 4, 7, 10, 14 and 21 for determination of ceftobiprole concentration in plasma. Safety evaluations including physical examination, vital signs, clinical laboratory tests, electrocardiogram and adverse event monitoring will be performed throughout the study. 500 mg ceftobiprole, intravenous infusion over 120 minutes, every 8 hours for 7 consecutive days

ELIGIBILITY:
Inclusion Criteria:

- Healthy volunteers with body weight >= 50 kg and body mass index between 18 and 30

* Agree to remain hospitalized at the trial unit during the 7-day drug administration period and will only leave the trial unit under supervision of a study nurse twice a day for one hour maximum
* Refrain from excessive jogging and any strenuous exercise during the study
* Be able to adhere to the dietary, fluid and smoking restrictions during the study
* Have negative pregnancy test result at the screening and agree to use adequate contraception method and not to become pregnant or donate sperm throughout the study

Exclusion Criteria:

* No clinically significant medical illness, abnormal findings in physical examination, vital signs, laboratory tests and electrocardiogram, or known allergy to the study drug, cephalosporins, beta-lactam antibiotics or other clinically significant allergies requiring treatment
* No antibiotic treatment within the last 3 months
* No drug or alcohol abuse within the last 5 years
* No blood donation or substantial loss of blood of more than 500 ml within the last 3 months or intention to donate blood during the study or within 1 month after study completion
* No history of smoking of more than 10 cigarettes , or 2 cigars, or 2 pipes of tobacco or 5 sniffs per day within the last 3 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Bacterial strains and numbers in feces; Minimum inhibitory concentrations for ceftobiprole for isolated resistant strains | Day 2, 4, 7, 10, 14 and 21

SECONDARY OUTCOMES:
Fecal concentration of ceftobiprole | Day 2, 4, 7, 10, 14 and 21
Plasma Concentration of ceftobiprole | Day 1, 4, 7, 10, 14, and 21

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV

REFERENCES:
- [Result] Backstrom T, Panagiotidis G, Beck O, Asker-Hagelberg C, Rashid MU, Weintraub A, Nord CE. Effect of ceftobiprole on the normal human intestinal microflora. Int J Antimicrob Agents. 2010 Dec;36(6):537-41. doi: 10.1016/j.ijantimicag.2010.07.021. PMID 20926263